CLINICAL TRIAL: NCT03615729
Title: RORC Genetic Polymorphism and Serum Levels in Patients With Rheumatoid Arthritis
Brief Title: RORC Genetic Polymorphism of Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Sayed, principal investigator, Assiut University
Other Study IDs: GPRA
Record Dates: First submitted 2018-07-22; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Genetic Predisposition to Disease
Keywords: Rheumatoid arthritis; Genetic polymorphism; RORc2 protein; T helper 17
MeSH Terms: conditions — Genetic Predisposition to Disease; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A total of 10 ml whole blood samples were obtained and were divided into two tubes; EDTA tube for genomic DNA extraction and serum-separating tubes for retinoic acid receptor-related orphan receptor variant 2 serum level determination by enzyme linked immunosorbant assay
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis patients: A total of 55 rheumatoid arthritis patients diagnosed according to 2010 ACR / EULAR Rheumatoid Arthritis Classification Criteria recruited from Clinical Rheumatology unit, Internal Medicine, Assiut University Hospitals
- controls: A total of 33 age and sex matched healthy controls randomly selected from healthy volunteers

SUMMARY:
Three candidate single nucleotide polymorphisms in the RORC2 gene, rs9826 A/G, rs3790515 C/T and rs3828057 C/T were examined together with estimation of nuclear hormone retinoic acid receptor-related orphan receptor variant 2 serum levels to determine their possible association with susceptibility to and clinical phenotype of rheumatoid arthritis in Egyptian population.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic systemic inflammatory arthritis that affects about one percent of the population. It results from a complex interaction between genes and environment (eg, external trigger as cigarette smoking, infection, or trauma) leading to a breakdown of immune tolerance, synovial inflammation and hypertrophy and chronic joint inflammation in a characteristic symmetric pattern.

The role of T helper 17 cells and T helper 17 cells -associated cytokines in the pathogenesis of rheumatoid arthritis is now widely recognized. T helper 17 cells are the dominant effector T cell involved in the induction of autoimmune chronic diseases by production of several proinflamatory cytokines especially interleukin -17. T helper 17 cells present in the joint may create a positive feedback loop leading to the continuous activation of T cells, which is a critical event in the generation of autoimmunity.

Nuclear hormone retinoic acid receptor-related orphan receptor variant 2, encoded by RORC2 gene located on chromosome 1q21-q23 is a master transcriptional factor that can drive T helper 17 cells differentiation. It is now well established that for T helper 17 cells differentiation, it is critical to have transforming growth factor β1 in the presence of interleukin-1, interleukin -6, or interleukin -21 to decrease suppressive FoxP3 and upregulate RORC2 gene encoded unique lineage-specific transcription factor, nuclear hormone retinoic acid receptor-related orphan receptor variant 2.

Knockdown of transcription factor nuclear hormone retinoic acid receptor-related orphan receptor variant 2 cause high forkhead transcriptional repressor levels and reduces expression of pro-inflammatory cytokines such as interleukin-1, interleukin -6, interleukin -17 and transforming growth factor β1 suggesting that the role of nuclear hormone retinoic acid receptor-related orphan receptor variant 2 in T helper 17 cells differentiation involves not only in induction of T helper 17 cells characteristics genes, but also suppression of Treg cells specific programs that play an important role in immunological tolerance.

Single nucleotide polymorphisms underlie differences in our susceptibility to disease, the severity of illness and the way our body responds to pathogens, chemicals, drugs, vaccines and other agents. For example, a single base mutation in the apolipoprotein E gene is associated with a higher risk for Alzheimer's disease.

RORC2 gene may represent a candidate gene for autoimmune diseases. However, not too much is known about the function of RORC2 genetic polymorphisms in autoimmune diseases, including rheumatoid arthritis. The RORC2 gene polymorphisms have been analyzed in a Behcet's disease, secondary lymphedema and type 2 diabetes mellitus and rheumatoid arthritis in a study on Polish population.

This is why analysis of polymorphisms within the RORC2 gene together with estimation of nuclear hormone retinoic acid receptor-related orphan receptor variant 2 serum levels may help to uncover their correlations with some clinical and laboratory findings in rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:- patients with rheumatoid arthritis diagnosed according to 2010 ACR / EULAR Rheumatoid Arthritis Classification Criteria

Exclusion Criteria:

1. Patients with other connective tissue diseases [e.g. systemic lupus erythematosis , systemic sclerosis, Behcet's disease,…etc]
2. Patients with other autoimmune diseases,
3. Patients with genetic diseases were excluded from the study
4. Patients with chronic liver or kidney diseases, . -

Ages: 20 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 55 patients (with rheumatoid arthritis diagnosed according to 2010 ACR / EULAR Rheumatoid Arthritis Classification Criteria) were recruited from Clinical Rheumatology unit, Internal Medicine, Assiut University Hospitals and 34 healthy volunteers were included in the study. Age of both of patients and healthy controls are 45.13 ± 10.6 years with a median age 45 years (20-73 years) and 43.00 ± 11.1 years with a median age 43 years (20-65 years) respectively. The numbers of females and males in RA patients are 50 and 5, respectively, and those in controls are 31 and 3 respectively.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Detection of SNPs genetic polymorphisms in RORC gene in rheumatoid arthritis | 2 hours
  Taqman SNP genotyping of rs9826 A/G, rs3790515 C/T and rs3828057 C/T in rheumatoid arthritis patients and control group to detect any possible association between RORC genetic polymorphism and rheumatoid arthritis

SECONDARY OUTCOMES:
Determination of serum Levels of RORc2 | 3 hours
  Determination of serum Levels of RORc2 were determined by enzyme-linked immunosorbent assay in rheumatoid arthritis patient and controls to determine RORc2 association with the risk and severity of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Hassanein, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikeda S, Saijo S, Murayama MA, Shimizu K, Akitsu A, Iwakura Y. Excess IL-1 signaling enhances the development of Th17 cells by downregulating TGF-beta-induced Foxp3 expression. J Immunol. 2014 Feb 15;192(4):1449-58. doi: 10.4049/jimmunol.1300387. Epub 2014 Jan 15. PMID 24431229
- [Background] Lee DM, Weinblatt ME. Rheumatoid arthritis. Lancet. 2001 Sep 15;358(9285):903-11. doi: 10.1016/S0140-6736(01)06075-5. PMID 11567728
- [Background] Liao D, Hou S, Zhang J, Fang J, Liu Y, Bai L, Cao Q, Kijlstra A, Yang P. Copy number variants and genetic polymorphisms in TBX21, GATA3, Rorc, Foxp3 and susceptibility to Behcet's disease and Vogt-Koyanagi-Harada syndrome. Sci Rep. 2015 Apr 15;5:9511. doi: 10.1038/srep09511. PMID 25873156
- [Background] Lim HW, Kang SG, Ryu JK, Schilling B, Fei M, Lee IS, Kehasse A, Shirakawa K, Yokoyama M, Schnolzer M, Kasler HG, Kwon HS, Gibson BW, Sato H, Akassoglou K, Xiao C, Littman DR, Ott M, Verdin E. SIRT1 deacetylates RORgammat and enhances Th17 cell generation. J Exp Med. 2015 May 4;212(5):607-17. doi: 10.1084/jem.20132378. Epub 2015 Apr 27. PMID 25918343
- [Background] Liu HP, Cao AT, Feng T, Li Q, Zhang W, Yao S, Dann SM, Elson CO, Cong Y. TGF-beta converts Th1 cells into Th17 cells through stimulation of Runx1 expression. Eur J Immunol. 2015 Apr;45(4):1010-8. doi: 10.1002/eji.201444726. Epub 2015 Feb 11. PMID 25605286
- [Background] Tesmer LA, Lundy SK, Sarkar S, Fox DA. Th17 cells in human disease. Immunol Rev. 2008 Jun;223:87-113. doi: 10.1111/j.1600-065X.2008.00628.x. PMID 18613831
- [Background] Wolf AB, Caselli RJ, Reiman EM, Valla J. APOE and neuroenergetics: an emerging paradigm in Alzheimer's disease. Neurobiol Aging. 2013 Apr;34(4):1007-17. doi: 10.1016/j.neurobiolaging.2012.10.011. Epub 2012 Nov 16. PMID 23159550
- [Background] Paradowska-Gorycka A, Stypinska B, Pawlik A, Romanowska-Prochnicka K, Haladyj E, Manczak M, Olesinska M. RORC2 Genetic Variants and Serum Levels in Patients with Rheumatoid Arthritis. Int J Mol Sci. 2016 Apr 1;17(4):488. doi: 10.3390/ijms17040488. PMID 27043554